CLINICAL TRIAL: NCT03115697
Title: High Volume Plasmapheresis for Refractory Hepatic Encephalopathy in Liver Intensive Care Unit-A Randomized Controlled Trial
Brief Title: High Volume Plasmapheresis for Refractory Hepatic Encephalopathy in Liver Intensive Care Unit.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HE-01
Record Dates: First submitted 2017-04-12; First posted 2017-04-14 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Refractory Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose; Rifaximin; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactulose with Rifaximin (Active Comparator)
  Interventions: Drug: Lactulose; Drug: Rifaximin
- Plasmapheresis (Experimental): Plasmapheresis will be added to the standard medical care therapy.(Maximum of 3 sessions once in 24 hours/or alternate days with an follow up for 5 days)
  Interventions: Biological: Plasmapheresis

INTERVENTIONS:
Drug: Lactulose — Lactulose 20 mL
  Arms: Lactulose with Rifaximin
Drug: Rifaximin — Rifaximin 550 BD
  Arms: Lactulose with Rifaximin
Biological: Plasmapheresis — Plasmapheresis 8 hrly duration
  Arms: Plasmapheresis

SUMMARY:
Study Design- Randomized Controlled trial Duration of enrolment-Feb-2016 to December 2017 Sample size-120 patients Methodology We will include consecutive with advanced hepatic encephalopathy not responding to treatment of precipitants and on treatment with Lactulose and Rifaximin for 48 hours .

Two groups will be divided. One arm -Lactulose and Rifaximin will be continued Second Arm - Plasmapheresis will be added to the standard medical care therapy.(Maximum of 3 sessions once in 24 hours/or alternate days with an follow up for 5 days)

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotics
* Age between 18-70 years
* Hepatic encephalopathy -Grade 3-4
* Patients receiving Lactulose/Rifaximin for 48 hours and not showing improvement in Hepatic encephalopathy(Persistent Grade 3/4)

Exclusion Criteria:

* Concomitant participation in an other clinical trial
* Patient receiving sedatives(propofol,etc) 24 hours prior.
* Patients with severe cardiopulmonary disease
* Pregnancy
* Human Immunodeficiency Virus
* Hepatocellular Carcinoma or extrahepatic malignancy
* Active uncontrolled sepsis with hemodynamic instability
* Chronic renal insufficiency on treatment with haemodialysis
* Uncontrolled bleed or patients in DIC
* Extremely moribund patients with expected survival of less than 48 hours on high vasopressor support
* Patients with moderate-severe Acute Respiratory Distress Syndrome (ARDS).
* Patients with Non Hepatic Coma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
Resolution in Hepatic Encephalopathy by 2 grades in both groups | Day 5

SECONDARY OUTCOMES:
Improvement in Hepatic Encephalopathy in both groups | 2 years
Number of days of mechanical ventilation in both groups | 2 years
Survival in both groups | 28 days
Proportion of patients with Systemic inflammatory response syndrome (SIRS) or sepsis as precipitants of Hepatic encephalopathy in both groups. | 2 years
Proportion of patients with failure of standard medical therapy in both groups. | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided